CLINICAL TRIAL: NCT04947709
Title: Physical Activity Post-Cancer for Adolescents and Young Adults (PAPAYA)
Brief Title: Physical Activity Post-Cancer for Adolescents and Young Adults
Acronym: PAPAYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Four Diamonds Research Fund at Penn State Health Childrens Hospital (Unknown)
Responsible Party: Principal Investigator, Smita Dandekar, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00018148
Record Dates: First submitted 2021-06-09; First posted 2021-07-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Childhood Cancer Survivors
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, utilizing a delayed-intervention control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity intervention group (Experimental): The physical activity intervention will be structured to increase moderate-to-vigorous intensity aerobic physical activity, to achieve the 60-minute goal, five days per week. The intervention will also include weekly support calls from research staff to improve compliance to physical activity intervention.
  Interventions: Behavioral: Physical Activity
- Delayed-intervention control group (Other): Participants randomized to the delayed-intervention control group will serve as the control group for 12 weeks, and will not receive physical activity intervention during this time and will not receive weekly support calls. After completion of the control group, participants will be offered physical activity advice according to the Children's Oncology Group Guidelines for Diet and Physical Activity recommendations. This delayed-intervention control group design is used not only to boost recruitment, but to eventually confer the benefits of physical activity to all those who enter the trial.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — The main structure of the physical activity program will focus on increasing physical activity. Physical activity will initially start at a duration of 15-30 minute bouts, and at rate of perceived exertion levels of 5-6 (somewhat hard). Over the course of the intervention, goals will be set to progress to 60 minutes of continuous physical activity, at a rate of perceived exertion level of 5-6 (somewhat hard). Participants will be instructed on the use of the ratings of the perceived exertion scale (Borg's RPE 1-10 scale). Participants will be instructed to walk, or engage in other forms of leisure-time physical activity to achieve these goals (cycling, running, swimming, etc). As the adolescent and young adults' health and fitness status improve, frequency, intensity, and session duration will be modified accordingly during weekly support calls. Moreover, goals will be responsive to the most recent week's achieved minutes and rate of perceived exertion.

SUMMARY:
The Physical Activity Post-Cancer for Adolescents and Young Adults (PAPAYA) trial aims to carry out a pilot randomized controlled trial among 10-17 year-old adolescents and young adults, at least 1 year and up to 5 years post-cancer treatment. The trial will evaluate the effects of a 12 week physical activity intervention to improve patient reported outcomes and physical function, in comparison to a delayed-intervention control group.

DETAILED DESCRIPTION:
The investigators will recruit 40 adolescents and young adults at least 1 year, and up to 5 years post-cancer treatment, and randomize them (20 randomized to each condition) to either a 12-week physical activity intervention to improve patient-reported outcomes and physical function, or delayed-intervention control group.

Participants randomized to the intervention group: The physical activity intervention will be structured to increase moderate-to-vigorous intensity aerobic physical activity, to achieve the 60 minute goal, five days per week. The intervention will also include weekly support calls from research staff. The physical activity intervention will be individualized by research staff according to the adolescents and young adults' health status, results from the physical fitness assessment, and most recent week's achieved minutes. The physical activity intervention will be modified during weekly support calls with a study team member, including frequency, intensity, time, and type, to maximize adherence and compliance

Participants randomized to the delayed-intervention control group: They will not receive the physical activity intervention, and they will not receive weekly support calls. Physical activity advice according to the Children's Oncology Group Guidelines for Diet and Physical Activity recommendations will be offered to participants randomized to the delayed-intervention control group following completion of 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

Adolescent and young adult inclusion criteria will be as follows:

1. males and females diagnosed with cancer;
2. treated at Penn State Health Children's Hospital or Penn State Cancer Institute, Milton S. Hershey Medical Center;
3. at least 1 year and up to 5 years post-cancer treatment;
4. being aged between 10 to 17 years old at enrollment;
5. being able to speak, read and understand the English language;
6. adolescents and young adults have to be able to assent, and parents/guardians have to be able to consent to the study in an informed manner;
7. Parent fluency in written and spoken English;
8. Adolescents and young adults or their parents must have access to a phone or Zoom

Note: The agreement of the attending oncologist will be required for the participation of adolescents and young adults eligible for this study.

Exclusion Criteria:

Adolescent and young adult exclusion criteria will be as follows:

1. Received follow-up at a location other than Penn State Health Children's Hospital or Penn State Cancer Institute, Milton S. Hershey Medical Center;
2. Evidence in the medical record of an absolute contraindication for physical activity;
3. cardiac exclusion criteria: Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system, history of acute coronary syndromes, uncertain or uncontrolled arrhythmia, uncontrolled hypertension, syncope, acute myocarditis, pericarditis, or endocarditis, acute pulmonary embolus or pulmonary infarction, thrombosis of lower extremities, suspected dissecting aneurysm, pulmonary edema, respiratory failure, acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise, mental impairment leading to inability to cooperate;
4. History of refractory or recurrent diseases
5. Already meeting physical activity guidelines.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Acceptability-the proportion of adolescents and young adults who agree to participate | Baseline
  The proportion of adolescents and young adults who agree to participate among those deemed eligible by the attending oncologist
  Range 0-100%-Higher scores indicate greater acceptability
Feasibility-the proportion of adolescents and young adults who complete at least 50% of the physical activity intervention | Baseline to week 12
  The percentage of those randomized to the physical activity intervention that complete at least 50% of the physical activity intervention. Participants will be instructed by a project manager during weekly support calls to accumulate a specific amount of physical activity each week. Participants who self-report completing at least 50% of the physical activity, determined by the Godin-Shephard Leisure-Time Physical Activity Questionnaire, will be deemed compliant.
  Range 0-100%-Higher scores indicate greater feasibility

SECONDARY OUTCOMES:
Patient reported outcomes-physical function mobility | Baseline
  the physical function mobility assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater physical function mobility
Patient reported outcomes-physical function mobility | week 12
  the physical function mobility assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater physical function mobility
Patient reported outcomes-anxiety | Baseline
  the anxiety assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater anxiety
Patient reported outcomes-anxiety | Week 12
  the anxiety assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater anxiety
Patient reported outcomes-depressive symptoms | baseline
  the depressive symptoms assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater depressive symptoms
Patient reported outcomes-depressive symptoms | Week 12
  the depressive symptoms assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater depressive symptoms
Patient reported outcomes-fatigue | baseline
  the fatigue assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater fatigue
Patient reported outcomes-fatigue | week 12
  the fatigue assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater fatigue
Patient reported outcomes-peer relationships | baseline
  the peer relationships assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater peer relationships
Patient reported outcomes-peer relationships | week 12
  the peer relationships assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater peer relationships
Patient reported outcomes-social isolation | baseline
  the social isolation assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater social isolation
Patient reported outcomes-social isolation | week 12
  the social isolation assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater social isolation
Patient reported outcomes-pain interference | baseline
  the pain interference assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater pain interference
Patient reported outcomes-pain interference | week 12
  the pain interference assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater pain interference
Patient reported outcomes-pain intensity | baseline
  the pain intensity assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 0-10, higher scores indicate greater pain intensity
Patient reported outcomes-pain intensity | week 12
  the pain intensity assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 0-10, higher scores indicate greater pain intensity
Patient reported outcomes-sleep disturbance | baseline
  the sleep disturbance assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater sleep disturbance
Patient reported outcomes-sleep disturbance | week 12
  the sleep disturbance assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 8-40, higher scores indicate greater sleep disturbance
Patient reported outcomes-cognitive function | baseline
  the cognitive function assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 7-35, higher scores indicate greater cognitive function
Patient reported outcomes-cognitive function | week 12
  the cognitive function assessment domain from the PROMIS (Patient-Reported Outcomes Measurement Information System Pediatric Profile v2.0-Profile-49)
  Range 7-35, higher scores indicate greater cognitive function
physical function-six minute walking test | baseline
  The six minute walking test will be administered to assess physical function. Participants will aim to walk as far as possible for 6 minutes.
  Further distances indicate greater physical function
physical function-six minute walking test | week 12
  The six minute walking test will be administered to assess physical function. Participants will aim to walk as far as possible for 6 minutes.
  Further distances indicate greater physical function
physical function-30 second chair stand | baseline
  The 30 second chair stand test will be administered to assess physical function. Participants will aim to sit and rise out of a chair as many times as possible in 30 seconds.
  Greater amounts of sit/stands indicate greater physical function
physical function-30 second chair stand | week 12
  The 30 second chair stand test will be administered to assess physical function. Participants will aim to sit and rise out of a chair as many times as possible in 30 seconds.
  Greater amounts of sit/stands indicate greater physical function
physical function-timed up and go | baseline
  The timed up and go test will be administered to assess physical function. Participants will aim to stand up, walk 3 meters, turn around, and walk back to the chair as fast as possible.
  Shorter durations indicate greater physical function
physical function-timed up and go | week 12
  The timed up and go test will be administered to assess physical function. Participants will aim to stand up, walk 3 meters, turn around, and walk back to the chair as fast as possible.
  Shorter durations indicate greater physical function

OTHER OUTCOMES:
Costs | Baseline to week 12
  Cost of carrying out the intervention will be also a secondary endpoint. We will include staff time, space, and equipment in our estimation of cost per patient to carry out the intervention
Demographics | baseline
  At baseline, assented/consented adolescents and young adults will be asked to complete the demographic questionnaires about age (years), sex (male or female), ethnicity (white or black or Asian or Hispanic other/mixed), education level. Adolescents and young adult participants will also be asked age at diagnosis (years), time since diagnosis (months) and diagnosis. Also, treatment interventions including cranial radiation (yes or no) and chemotherapy (yes or no) will be obtained. Adolescents and young adults will be asked if they are currently receiving any mental health-related treatment and/or intervention.
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | Baseline
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 1
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 2
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 3
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 4
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 5
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 6
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 7
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 8
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 9
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 10
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 11
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Physical activity-Godin-Shephard Leisure-Time Physical Activity Questionnaire (process outcome) | week 12
  Physical activity will be assessed by a self-reported, 4-item questionnaire. This questionnaire will be administered over the telephone or HIPAA compliant ZOOM weekly. Weekly frequencies of strenuous, moderate, and light activities are reported, and using a standardized formula, total weekly leisure activity is calculated.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active

CONTACTS AND LOCATIONS:
Overall Officials: Smita Dandekar, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Caru M, Dandekar S, Gordon B, Conroy DE, Barb ED, Doerksen SE, Smink GM, McKeone DJ, Shah NB, Greiner RJ, Schramm JW, Rao P, McGregor L, Schmitz KH. Implementing a behavioral physical activity program in children and adolescent survivors of childhood cancer: a pilot randomized controlled trial. J Behav Med. 2024 Oct;47(5):792-803. doi: 10.1007/s10865-024-00497-z. Epub 2024 May 12. PMID 38735024